CLINICAL TRIAL: NCT06575205
Title: A Brief Patient Educational Video to Reduce Potentially Harmful Over-the-counter Nonsteroidal Anti-inflammatory Drug (NSAID) Use
Brief Title: Patient Education Video to Reduce OTC NSAIDs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Michelle Rockwell, Assistant Professor, Principal Investigator, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-22-1766
Record Dates: First submitted 2023-08-14; First posted 2024-08-28 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Heart Failure; Hypertension
Keywords: Chronic Kidney Diseases; Heart Failure; Hypertension; Over the Counter NSAIDS
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure; Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): An original brief 3 to 5 minute educational video, covering themes such as: defining OTC NSAIDs and their uses, potential harms of NSAIDs, and broad general alternatives. Will involve suggestion to speak to their healthcare provider.
  Interventions: Behavioral: Educational video
- Control (No Intervention): A static image of a standardized FDA warning label for OTC NSAIDs covering themes such as: uses of OTC NSAIDs, potential harms of NSAIDs, and suggestion to speak to their healthcare provider.

INTERVENTIONS:
Behavioral: Educational video — Participants will view a brief 3-to-5-minute educational video (VIDEO), covering information that is already printed on FDA labels for OTC NSAIDs, on their own device covering themes such as: defining OTC NSAIDs, potential harms of NSAIDs, and alternatives.
  Arms: Video

SUMMARY:
The goal of this study is to assess the efficacy of a brief 3 to 5-minute educational video on influencing intent to change behavior regarding potentially harmful over-the-counter (OTC) NSAID use in adults with chronic kidney disease (CKD), heart failure (HF), and/or hypertension (HTN). Informed by the COM-B model of behavior change, the video reviews identifying OTC NSAIDs, potential risks of NSAIDs, and general alternatives to potentially harmful NSAIDs. Participants with CKD, HF, and/or HTN identified as regular OTC NSAID users will be randomized to the VIDEO or CONTROL group. They will complete surveys immediately and 4 weeks after viewing the VIDEO or CONTROL to assess actual NSAIDs use, intent to change behavior related to NSAIDs use, capability/opportunity/motivation to change behavior, pain, and barriers to decreasing OTC NSAIDs. Findings will inform future population health initiatives to reduce potentially harmful OTC NSAIDs use.

DETAILED DESCRIPTION:
Nonsteroidal anti-inflammatory drugs (NSAIDs) are effective in treating pain and inflammation, but are also associated with multiple risks for some patients. Numerous organizations recommend that older adults and patients with chronic diseases such as kidney disease, heart failure, and hypertension avoid chronic use of NSAIDs. However, high-risk use persists at undesirable rates. The goal of this study is to assess the efficacy of an original, brief, 3 to 5 minute educational video, on influencing intent to change behavior regarding potentially harmful over-the-counter (OTC) NSAID use. The study population will involve adult patients from a large regional health system in the southeastern U.S. with a diagnosis of chronic kidney disease (CKD), heart failure (HF), and/or hypertension (HTN) as NSAID use is contraindicated in this population.

All patients with a diagnosis of CKD, HF, and/or HTN, who have an email address on file will be invited to participate via email/REDCap. Upon clicking the link, general study information will be provided for participant informed consent and a printable IRB subject informational sheet will be made available to all potential participants and participants. After acknowledgment by the participant, a pre-educational survey will assess recent use of over-the-counter NSAIDs and general demographic information. Those who meet criteria for regular NSAIDs use (>3 doses per week over previous 3 months) will be immediately invited to participate in a randomized controlled trial (Education Tool Survey accompanied by VIDEO or CONTROL).

Participants will answer 3 additional baseline pain level survey questions and 1 additional question regarding their baseline intent to change their current use of OTC NSAIDs. Participants will then immediately be randomized to either view the brief 3 to 5 minute educational video (VIDEO) on their own device covering themes that are already covered on the FDA warning label such as: defining OTC NSAIDs, potential harms of NSAIDs, and alternatives or participants will view a standard OTC NSAIDs FDA warning label (CONTROL). Trial participants will complete a survey electronically immediately after viewing VIDEO or CONTROL covering questions about intent to change behaviors related to OTC NSAID use and barriers, capability, opportunity, and motivation to change behaviors. This portion of the study will take less than 10 minutes to complete.

Trial participants will complete a survey electronically again 4 weeks later regarding questions about intent to change the use of OTC NSAIDs, actual use of OTC NSAIDs (for the recent 4 week time period), levels of pain, and barriers, capability, opportunity, and motivation to change behaviors. REDCap will auto-send the 4 week survey 4 weeks after completion of the Education Tool Survey. This portion of the study will take less than 5 minutes to complete.

The study team will perform a multivariable linear regression to evaluate the association of demographics on OTC NSAID use. The study team will use paired t-tests to evaluate group and time differences. The study team will use stepwise forward multivariable linear regression to evaluate the relative impact of secondary outcomes (barriers, capability, opportunity, and motivation to change behaviors, and ratings of pain) on intent to change NSAID use. Spearman's correlation analysis will also be performed between all variables. Significance will be set at the 0.05 level.

Results of this study will inform population health interventions to reduce potentially harmful OTC NSAIDs use.

ELIGIBILITY:
Inclusion Criteria:

* Carilion Clinic patients
* Age > = 18 years
* Diagnosis of CKD, HTN, and/or HF
* E-mail address or phone number on file.
* Able to speak and read English
* Able to respond to an online survey and view a video

Exclusion Criteria:

* Not Carilion Clinic patients
* Age < 18
* No diagnosis of CKD, HTN, or HF
* No e-mail address or phone number on file
* Cannot speak or read English
* Not able to respond to an online survey or view a video

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Contemplation Ladder score | baseline prior to viewing VIDEO or CONTROL and within 10 minutes after viewing VIDEO or CONTROL and 4 weeks later
  Intent to change behavior related to OTC NSAID use, scored from 0 (no intent to decrease OTC NSAID use) to 10 (already committed to decreasing OTC NSAID use). A higher score is the better outcome (greater intent to decrease high-risk OTC NSAIDs).
Self-reported OTC NSAID use | baseline prior to viewing VIDEO or CONTROL and 4 weeks later
  NSAID use over the past 30 days, reported as number of days during the past 30 that OTC NSAIDs were used. The range of responses is 0 to 30.

SECONDARY OUTCOMES:
Barriers to decreasing OTC NSAIDs use | baseline prior to viewing VIDEO or CONTROL and 4 weeks later
  Participant response to open-ended survey question: What is the biggest barrier to decreasing your use of OTC NSAIDs?
Capability to decrease OTC NSAIDs use score | baseline prior to viewing VIDEO or CONTROL and 4 weeks later
  2 survey questions focused on capability portion of COM-B model of behavior change. This question is scored on an 11-point likert scale, from 0 to 11. A score of 11 indicates the greatest perceived capability.
Motivation to decrease OTC NSAIDs use score | baseline prior to viewing VIDEO or CONTROL and 4 weeks later
  2 survey questions focused on motivation portion of COM-B model of behavior change. This question is scored on an 11-point likert scale, from 0 to 11. A score of 11 indicates the greatest perceived motivation.
Rating of pain score | baseline prior to viewing VIDEO or CONTROL and 4 weeks later
  Response to question: rate your pain over the past 30 days. This will be scored on a 6-point likert scale with 0=no pain and 5=severe pain.
Opportunity to decrease OTC NSAIDs use score | baseline prior to viewing VIDEO or CONTROL and 4 weeks later
  2 survey questions focused on opportunity portion of COM-B model of behavior change. This question is scored on an 11-point likert scale, from 0 to 11. A score of 11 indicates the greatest perceived opportunity.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Rockwell, PhD, RD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic Riverside 1, Roanoke, Virginia, United States

REFERENCES:
- [Background] Antman EM, Bennett JS, Daugherty A, Furberg C, Roberts H, Taubert KA; American Heart Association. Use of nonsteroidal antiinflammatory drugs: an update for clinicians: a scientific statement from the American Heart Association. Circulation. 2007 Mar 27;115(12):1634-42. doi: 10.1161/CIRCULATIONAHA.106.181424. Epub 2007 Feb 26. No abstract available. PMID 17325246
- [Background] Arfe A, Scotti L, Varas-Lorenzo C, Nicotra F, Zambon A, Kollhorst B, Schink T, Garbe E, Herings R, Straatman H, Schade R, Villa M, Lucchi S, Valkhoff V, Romio S, Thiessard F, Schuemie M, Pariente A, Sturkenboom M, Corrao G; Safety of Non-steroidal Anti-inflammatory Drugs (SOS) Project Consortium. Non-steroidal anti-inflammatory drugs and risk of heart failure in four European countries: nested case-control study. BMJ. 2016 Sep 28;354:i4857. doi: 10.1136/bmj.i4857. PMID 27682515
- [Background] Coxib and traditional NSAID Trialists' (CNT) Collaboration; Bhala N, Emberson J, Merhi A, Abramson S, Arber N, Baron JA, Bombardier C, Cannon C, Farkouh ME, FitzGerald GA, Goss P, Halls H, Hawk E, Hawkey C, Hennekens C, Hochberg M, Holland LE, Kearney PM, Laine L, Lanas A, Lance P, Laupacis A, Oates J, Patrono C, Schnitzer TJ, Solomon S, Tugwell P, Wilson K, Wittes J, Baigent C. Vascular and upper gastrointestinal effects of non-steroidal anti-inflammatory drugs: meta-analyses of individual participant data from randomised trials. Lancet. 2013 Aug 31;382(9894):769-79. doi: 10.1016/S0140-6736(13)60900-9. Epub 2013 May 30. PMID 23726390
- [Background] Choosing Wisely American Society of Nephrology NSAIDs Recommendation. https://www.choosingwisely.org/clinician-lists/american-society-nephrology-nsaids-in-individuals-with-hypertension-heart-failure-or-chronic-kidney-disease/, accessed March 2022
- [Background] Davis JS, Lee HY, Kim J, Advani SM, Peng HL, Banfield E, Hawk ET, Chang S, Frazier-Wood AC. Use of non-steroidal anti-inflammatory drugs in US adults: changes over time and by demographic. Open Heart. 2017 Apr 28;4(1):e000550. doi: 10.1136/openhrt-2016-000550. eCollection 2017. PMID 28674622
- [Background] Davison SN, Koncicki H, Brennan F. Pain in chronic kidney disease: a scoping review. Semin Dial. 2014 Mar;27(2):188-204. doi: 10.1111/sdi.12196. Epub 2014 Feb 12. PMID 24517512
- [Background] Gates, B. J., Setter, S. M., Corbett, C. F., & Baker, D. E. (2005). A Comparison of Educational Methods to Improve NSAID Knowledge and Use of a Medication List in an Elderly Population. Home Health Care Management & Practice, 17(5), 403-410.
- [Background] Green GA. Understanding NSAIDs: from aspirin to COX-2. Clin Cornerstone. 2001;3(5):50-60. doi: 10.1016/s1098-3597(01)90069-9. PMID 11464731
- [Background] Hales CM, Martin CB, Gu Q. Prevalence of Prescription Pain Medication Use Among Adults: United States, 2015-2018. NCHS Data Brief. 2020 Jun;(369):1-8. PMID 32600518
- [Background] Harirforoosh S, Asghar W, Jamali F. Adverse effects of nonsteroidal antiinflammatory drugs: an update of gastrointestinal, cardiovascular and renal complications. J Pharm Pharm Sci. 2013;16(5):821-47. doi: 10.18433/j3vw2f. PMID 24393558
- [Background] Koffeman AR, Valkhoff VE, Celik S, W't Jong G, Sturkenboom MC, Bindels PJ, van der Lei J, Luijsterburg PA, Bierma-Zeinstra SM. High-risk use of over-the-counter non-steroidal anti-inflammatory drugs: a population-based cross-sectional study. Br J Gen Pract. 2014 Apr;64(621):e191-8. doi: 10.3399/bjgp14X677815. PMID 24686883
- [Background] Labelle M, Beaulieu M, Paquette D, Fournier C, Bessette L, Choquette D, Rahme E, Thivierge RL. An integrated approach to improving appropriate use of anti-inflammatory medication in the treatment of osteoarthritis in Quebec (Canada): the CURATA model. Med Teach. 2004 Aug;26(5):463-70. doi: 10.1080/0142159042000218669. PMID 15369888
- [Background] Lefebvre C, Hindie J, Zappitelli M, Platt RW, Filion KB. Non-steroidal anti-inflammatory drugs in chronic kidney disease: a systematic review of prescription practices and use in primary care. Clin Kidney J. 2019 May 20;13(1):63-71. doi: 10.1093/ckj/sfz054. eCollection 2020 Feb. PMID 32082554
- [Background] Martin P, Tamblyn R, Benedetti A, Ahmed S, Tannenbaum C. Effect of a Pharmacist-Led Educational Intervention on Inappropriate Medication Prescriptions in Older Adults: The D-PRESCRIBE Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1889-1898. doi: 10.1001/jama.2018.16131. PMID 30422193
- [Background] McDonald DD, Amendola MG, Interlandi E, Wall K, Lewchik B, Polouse L, Pace N, Inthavong S, Li L. Effect of reading additional safety information on planned use of over-the-counter analgesics. Public Health Nurs. 2007 May-Jun;24(3):230-8. doi: 10.1111/j.1525-1446.2007.00629.x. PMID 17456124
- [Background] Morrison C, Beauchamp T, MacDonald H, Beattie M. Implementing a non-steroidal anti-inflammatory drugs communication bundle in remote and rural pharmacies and dispensing practices. BMJ Open Qual. 2018 Jul 21;7(3):e000303. doi: 10.1136/bmjoq-2017-000303. eCollection 2018. PMID 30057956
- [Background] Mullan J, Weston KM, Bonney A, Burns P, Mullan J, Rudd R. Consumer knowledge about over-the-counter NSAIDs: they don't know what they don't know. Aust N Z J Public Health. 2017 Apr;41(2):210-214. doi: 10.1111/1753-6405.12589. Epub 2016 Oct 24. PMID 27774735
- [Background] National Kidney Foundation. Pain Medicine and Your Kidneys. https://www.kidney.org/atoz/content/painmeds_analgesics. Accessed March 2022
- [Background] Neafsey PJ, M'lan CE, Ge M, Walsh SJ, Lin CA, Anderson E. Reducing Adverse Self-Medication Behaviors in Older Adults with Hypertension: Results of an e-health Clinical Efficacy Trial. Ageing Int. 2011 Jun;36(2):159-191. doi: 10.1007/s12126-010-9085-9. Epub 2010 Dec 8. PMID 21654869
- [Background] Pandolfe F, Crotty BH, Safran C. Medication Harmony: A Framework to Save Time, Improve Accuracy and Increase Patient Activation. AMIA Annu Symp Proc. 2017 Feb 10;2016:1959-1966. eCollection 2016. PMID 28269955
- [Background] Vane JR, Botting RM. Anti-inflammatory drugs and their mechanism of action. Inflamm Res. 1998 Oct;47 Suppl 2:S78-87. doi: 10.1007/s000110050284. PMID 9831328
- [Background] Ungprasert P, Cheungpasitporn W, Crowson CS, Matteson EL. Individual non-steroidal anti-inflammatory drugs and risk of acute kidney injury: A systematic review and meta-analysis of observational studies. Eur J Intern Med. 2015 May;26(4):285-91. doi: 10.1016/j.ejim.2015.03.008. Epub 2015 Apr 8. PMID 25862494
- [Background] U.S. Food and Drug Administration. Acetaminophen overdose and liver injury- background and options for reducing injury. (2011) http://www.fda.gov/downloads/ AdvisoryCommittees/CommitteesMeetingMaterials/Drugs/DrugSafetyandRisk ManagementAdvisoryCommittee/UCM164897.pdf (accessed April 27, 2022).
- [Background] Wehling M. Non-steroidal anti-inflammatory drug use in chronic pain conditions with special emphasis on the elderly and patients with relevant comorbidities: management and mitigation of risks and adverse effects. Eur J Clin Pharmacol. 2014 Oct;70(10):1159-72. doi: 10.1007/s00228-014-1734-6. Epub 2014 Aug 28. PMID 25163793
- [Background] Whelton A. Nephrotoxicity of nonsteroidal anti-inflammatory drugs: physiologic foundations and clinical implications. Am J Med. 1999 May 31;106(5B):13S-24S. doi: 10.1016/s0002-9343(99)00113-8. PMID 10390124
- [Background] Wilcox CM, Cryer B, Triadafilopoulos G. Patterns of use and public perception of over-the-counter pain relievers: focus on nonsteroidal antiinflammatory drugs. J Rheumatol. 2005 Nov;32(11):2218-24. PMID 16265706
- [Background] Wongrakpanich S, Wongrakpanich A, Melhado K, Rangaswami J. A Comprehensive Review of Non-Steroidal Anti-Inflammatory Drug Use in The Elderly. Aging Dis. 2018 Feb 1;9(1):143-150. doi: 10.14336/AD.2017.0306. eCollection 2018 Feb. PMID 29392089
- [Background] Zhan M, Doerfler RM, Xie D, Chen J, Chen HY, Diamantidis CJ, Rahman M, Ricardo AC, Sondheimer J, Strauss L, Wagner LA, Weir MR, Fink JC; CRIC Study Investigators. Association of Opioids and Nonsteroidal Anti-inflammatory Drugs With Outcomes in CKD: Findings From the CRIC (Chronic Renal Insufficiency Cohort) Study. Am J Kidney Dis. 2020 Aug;76(2):184-193. doi: 10.1053/j.ajkd.2019.12.010. Epub 2020 Apr 18. PMID 32317121
- [Background] Zhou Y, Boudreau DM, Freedman AN. Trends in the use of aspirin and nonsteroidal anti-inflammatory drugs in the general U.S. population. Pharmacoepidemiol Drug Saf. 2014 Jan;23(1):43-50. doi: 10.1002/pds.3463. Epub 2013 May 30. PMID 23723142